CLINICAL TRIAL: NCT01657942
Title: Focal MR-Guided Focused Ultrasound Treatment of Localized Intermediate Risk Prostate Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: InSightec (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PCa003
Record Dates: First submitted 2012-08-02; First posted 2012-08-06 (Estimated); Results first posted 2024-11-13 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-10

CONDITIONS: Localized Intermediate Risk Prostate Lesions
Keywords: MRgFUS; Prostate; Intermediate Risk Prostate Lesions; Focal Prostate treatment; InSightec; ExAblate; Non-invasive; Prostate cancer; Gleason 7
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ExABlate MR Guided Focus Ultrasound (Experimental): ExAblate MR Guided Focused Ultrasound - Local treatment of prostate lesions using Magnetic Resonance Imaging guided endorectally applied focused ultrasound energy.
  Interventions: Device: ExAblate MR Guided Focused Ultrasound

INTERVENTIONS:
Device: ExAblate MR Guided Focused Ultrasound — ExAblate MR Guided Focused Ultrasound - Local treatment of prostate lesions using Magnetic Resonance Imaging guided endorectally applied focused ultrasound energy.
  Other Names: ExAblate 2100 Prostate System

SUMMARY:
The hypothesis of this study is that focal treatment with ExAblate MRgFUS has the potential to be an effective non-invasive treatment for intermediate risk, organ-confined prostate lesions, with a low incidence of morbidity. The study hypothesis will be tested by measuring treatment-related safety and initial effectiveness parameters in the ExAblate MRgFUS treated patients, as described above.

DETAILED DESCRIPTION:
Objective of this pivotal trial is to assess safety and initial effectiveness of ExAblate MRgFUS in the treatment of intermediate risk, localized (organ confined) prostate lesions.

ExAblate treatment will be implemented as a focal lesion-selective therapy, directed at pre-defined volume(s)/sector(s) in the prostate, identified by mapping biopsy and multi-parametric MRI, rather than a whole gland or hemi-ablation treatment.

Safety: evaluate incidence and severity of adverse events associated with ExAblate's MRgFUS focal treatment of intermediate risk organ confined prostate lesions. The risk of ExAblate treatment-related incontinence and impotence will also be assessed in this study.

Effectiveness: determine the lesion control effect of ExAblate's MRgFUS focal treatment of intermediate risk organ-confined prostate lesions (confirmed by IMAGE-guided mapping biopsy results).

ELIGIBILITY:
Inclusion Criteria

* Biopsy proven adenocarcinoma of the prostate (using a IMAGE-guided 14+ core mapping biopsy), and targeted cores as needed obtained up to 6 months prior to scheduled treatment
* Patient with intermediate risk, early-stage organ-confined prostate cancer (T1a up to T2b, N0, M0) and voluntarily chooses ExAblate thermal ablation as the non-invasive treatment, who may currently be on watchful waiting or active surveillance and not in need of imminent radical therapy.
* Patient with PSA less than or equal to 20 ng/mL
* Gleason score 7 (4 + 3 or 3 + 4), based on mapping prostate biopsy, with no more than 15mm cancer in maximal linear dimension in any single core
* Single hemilateral index Gleason 7 lesion, identified in the prostate based on biopsy mapping with supporting MRI; may have secondary Gleason 6 lesion on ipsilateral or contralateral side confirmed with biopsy and/or MRI

Exclusion Criteria

* Contraindications to MRI
* History of orchiectomy, PCa-specific chemotherapy, brachytherapy, cryotherapy, Photodynamic therapy or radical prostatectomy for treatment of prostate cancer; any prior radiation therapy to the pelvis for prostate cancer or any other malignancy
* Patient under medications that can affect PSA for the last 3 months prior to MRgFUS treatment (Androgen Deprivation Treatment; alpha reductase inhibitors)
* Individuals who are not able or willing to tolerate the required prolonged stationary supine position during treatment (approximately 3 hrs. sonication time)
* Any rectal pathology, anomaly or previous treatment, which could change acoustic properties of rectal wall or prevent safe probe insertion (e.g., stenosis, fibrosis, inflammatory bowel disease, etc.)
* Evidence of distant prostate cancer, i.e., including lymph nodes and/or metastasis of cancer on imaging
* Bladder cancer
* Urethral stricture/bladder neck contracture
* Prostatitis NIH categories I, II and III
* Implant near (<1 cm) the prostate

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2019-10 (Actual); Study Completion 2021-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Behfar Ehdaie, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (9):
- United States (9):
  - City of Hope, Duarte, California
  - University of California Los Angeles, Los Angeles, California
  - Stanford University School of Medicine, Stanford, California
  - Sperling Prostate Center, Delray Beach, Florida
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Weill Cornell Medical Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - University of Virginia, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bitton RR, Shao W, Chodakeiwitz Y, Brunsing RL, Sonn G, Rusu M, Ghanouni P. Intraprocedural Diffusion-weighted Imaging for Predicting Ablation Zone during MRI-guided Focused Ultrasound of Prostate Cancer. Radiol Imaging Cancer. 2024 Sep;6(5):e240009. doi: 10.1148/rycan.240009. PMID 39212524
- [Derived] Ehdaie B, Tempany CM, Holland F, Sjoberg DD, Kibel AS, Trinh QD, Durack JC, Akin O, Vickers AJ, Scardino PT, Sperling D, Wong JYC, Yuh B, Woodrum DA, Mynderse LA, Raman SS, Pantuck AJ, Schiffman MH, McClure TD, Sonn GA, Ghanouni P. MRI-guided focused ultrasound focal therapy for patients with intermediate-risk prostate cancer: a phase 2b, multicentre study. Lancet Oncol. 2022 Jul;23(7):910-918. doi: 10.1016/S1470-2045(22)00251-0. Epub 2022 Jun 14. PMID 35714666

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was multi-center, prospective, single arm, observational trial conducted in the United States where subjects were treated and followed for 12 months. Males over 50 years of age (median age of 63 years) with a single, MRI-visible, hemilateral lesion of biopsy proven Gleason Grade Group 2 (3+4) or 3 (4+3) adenocarcinoma and with a PSA less than or equal to 20 ng/mL were treated with the Exablate 2100 Prostate System.
Groups:
- Exablate MR Guided Focus Ultrasound Treatment of Locally Confined Intermediate Risk Prostate Lesions: Single Arm Study: Exablate MR Guided Focused Ultrasound for local treatment of prostate lesions using Magnetic Resonance (MR) to guide focused ultrasound energy.
Period: Overall Study
Arm/Group | Exablate MR Guided Focus Ultrasound Treatment of Locally Confined Intermediate Risk Prostate Lesions
Started | 101
Post Treatment Assignment Group 1) Involvement of Neurovascular Bundles and/or Urethra | 57 (Post treatment results in terms of Patient-reported assessments were reported in two groups: 1) neurovascular bundles and/or urethra included in the treatment (n=57), or 2) neurovascular bundles and/or urethra NOT included in the treatment (n=44).)
Post Treatment Assignment Group 2) no Involvement of Neurovascular Bundles and/or Urethra | 44 (Post treatment results in terms of Patient-reported assessments were reported in two groups: 1) neurovascular bundles and/or urethra included in the treatment (n=57), or 2) neurovascular bundles and/or urethra NOT included in the treatment (n=44).)
Completed | 93
Not Completed | 8
Not completed — Alternative Treatment | 7
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Groups:
- Exablate MR Guided Focus Ultrasound Treatment of Localized Intermediate Risk Prostate Lesions: Exablate MR Guided Focused Ultrasound for the local treatment of intermediate prostate lesions using Magnetic Resonance guided focused ultrasound energy.
Arm/Group | Exablate MR Guided Focus Ultrasound Treatment of Localized Intermediate Risk Prostate Lesions
Number analyzed (Participants) | 101
Age, Continuous [Mean (Standard Deviation); unit: Years]
  Age | 62.9 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 101
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 90
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 101
Biopsy proven adenocarcinoma of the prostate [Count of Participants; unit: Participants] | 101
BMI [kg/m^2] [Mean (Standard Deviation); unit: kg/m^2] | 28.5 (4.5)
Weight [kg] [Mean (Standard Deviation); unit: kg] | 91.3 (17.3)

OUTCOME MEASURES:

1. Primary Outcome: Number of Device and Procedure Related Adverse Events
Description: The cumulative sum of adverse events was followed through Month 12 of the study.
Time Frame: 12 months Post Treatment
Population: Adverse Events and Serious Adverse Events are reported in the Adverse Events Section.
Measure: Number; unit: Number of Adverse Events
Groups:
- Exablate MR Guided Focus Ultrasound: Exablate MR Guided Focused Ultrasound - Local treatment of prostate lesions using Magnetic Resonance guided focused ultrasound energy
Arm/Group | Exablate MR Guided Focus Ultrasound
Number analyzed (Participants) | 101
Number of Adverse Events | 24

2. Primary Outcome: Percentage of Subjects With NO Gleason Grade Group (GGG) Tissue in the Planned Region of Treatment (ROT) at 6 Months.
Description: The first primary effectiveness endpoint is within area of treatment (Region of Treatment, ROT) prostate biopsy occurring at 6-months post-treatment. Positive biopsy was defined as any Gleason Grade Group (GGG) tissue identified within the area of planned Exablate ROT. Negative biopsy was defined No Gleason Grade Group (GGG) tissue within the area of planned ROT.
Time Frame: 6 Months Post Treatment
Measure: Number (95% Confidence Interval); unit: Percentage of Subjects
Groups:
- Exablate MR Guided Focused Ultrasound: Exablate MR Guided Focused Ultrasound for the local treatment of prostate lesions using Magnetic Resonance guided focused ultrasound energy
Arm/Group | Exablate MR Guided Focused Ultrasound
Number analyzed (Participants) | 101
Percentage of Subjects | 91.1 [83.8 to 95.8]

3. Primary Outcome: Percentage of Subjects Showing a Reduction in PSA Value (Prostate Specific Antigen) From Baseline to 6-Months
Description: The second primary effectiveness endpoint is the percentage of subjects experiencing a reduction in PSA value (Prostate Specific Antigen) from baseline to 6-months post-treatment. PSA values that increased or remained the same were considered an increase. Increased Prostate Specific Antigen levels in the blood is a common indication of prostate cancer.
  PSA results at 6 months - Value of ≤ 10ng/mL (Yes/No)
Time Frame: 6-months Post Treatment
Measure: Number (95% Confidence Interval); unit: Percentage of Subjects
Arm/Group | Exablate MR Guided Focus Ultrasound
Number analyzed (Participants) | 101
Percentage of Subjects | 91.1 [83.8 to 95.8]

4. Primary Outcome: Percentage of Subjects With Non-Perfused Volume (NPV) Entirely Covered Target Gleason Grade Group (GGG) Tissue at Treatment.
Description: The final primary effectiveness endpoint is percentage of subjects with NPV complete coverage of targeted Gleason tissue at treatment. NPV (non-perfused volume) is the volume of tissue ablated/treated, a measure of the completeness/effectiveness of the ablation.
Time Frame: 6 Months Post Treatment
Measure: Number (95% Confidence Interval); unit: Percentage of Subjects
Arm/Group | Exablate MR Guided Focus Ultrasound
Number analyzed (Participants) | 101
Percentage of Subjects | 87.1 [79.0 to 93.0]

5. Secondary Outcome: Prostate Specific Antigen (PSA)
Description: Prostate Specific Antigen (PSA) concentration in the blood is commonly measured to screen for prostate cancer. Prostate Specific Antigen (PSA) was reported as a primary endpoint. Here it is presented to show levels at 6 Months and 12 Months post-treatment compared to Baseline (pre-treatment). Elevated PSA suggests potential cancer.
Time Frame: Baseline, 6 Months, 12 Months
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Exablate MR Guided Focus Ultrasound
Number analyzed (Participants) | 101
ng/mL
  Baseline | 6.4 (3.1)
  6 Months | 3.3 (2.9)
  12 Months | 3.2 (2.5)

6. Secondary Outcome: Functional Assessment of Cancer Therapy - General (Fact-G) Total Score
Description: The total FACT-G score ranges from 0 to 108 and is the summation of 4 subscale scores. The subscale scores are added to obtain the total score, which is calculated using a five-point scale from 0 (not at all) to 4 (very much). A higher FACT-G score indicates better overall well-being and quality of life. The FACT-G is an alternative scoring method to the Trial Outcome Index (TOI) which is also reported in this study.
Time Frame: Baseline, 3 Months, 6 Months, 9 Months, 12 Months.
Population: Deviations across visits resulted from missed visits and missed assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Neurovascular Bundles and/or Urethra Included in Treatment: For patient self-completed assessents subjects were separated into two subgroups after the treatment (not randomly): 1) Neurovascular bundles and/or urethra included in treatment (n=57) or 2) Neurovascular bundles and urethra NOT included in treatment (n=44). There was no hypothesis test comparison between groups. Comparisons are only observational. Deviations from the Overall Number of Participants is a result of missed visits, assessments and early exits.
- Neurovascular Bundles and Urethra Not Included in Treatment: For patient self-completed assessents subjects were separated into two subgroups after the treatment (not randomly: 1) Neurovascular bundles and/or urethra included in treatment (n=57) or 2) Neurovascular bundles and urethra NOT included in treatment (n=44). There was no hypothesis test comparison between groups. Comparisons are only observational. Deviations from the Overall Number of Participants is a result of missed visits, assessments and early exits.
- Total Exablate MR Guided Focus Ultrasound: Combined Groups: Exablate MR Guided Focused Ultrasound - Local treatment of prostate lesions using Magnetic Resonance guided focused ultrasound energy. Combined groups (n=101): 1) Neurovascular bundles and/or urethra included in treatment (n=57) or 2) Neurovascular bundles and urethra NOT included in treatment (n=44).
Arm/Group | Neurovascular Bundles and/or Urethra Included in Treatment | Neurovascular Bundles and Urethra Not Included in Treatment | Total Exablate MR Guided Focus Ultrasound
Number analyzed (Participants) | 57 | 44 | 101
score on a scale
  Baseline | 94.8 (10.8) | 94.5 (8.8) | 94.7 (9.9)
  3 Months: number analyzed (Participants) | 56 | 44 | 100
  3 Months | 95.7 (8.5) | 90.2 (12.7) | 93.3 (10.9)
  6 Months: number analyzed (Participants) | 55 | 42 | 97
  6 Months | 64.0 (10.8) | 92.5 (11.0) | 93.4 (10.9)
  9 Months: number analyzed (Participants) | 50 | 38 | 88
  9 Months | 97.3 (7.7) | 92.3 (10.7) | 95.1 (9.4)
  12 Months: number analyzed (Participants) | 51 | 39 | 90
  12 Months | 95.3 (10.8) | 93.3 (10.5) | 94.4 (10.7)

7. Secondary Outcome: Functional Assessment of Cancer Therapy - Prostate (Fact P) Total Score
Description: The Fact-P Total Score (Score range: 0-156) is a comprehensive multidimensional quality of life measure designed specifically for patients with prostate cancer. It is a 39-item assessment in a 5-point (0-4) Likert-type Scale. Higher scores represent better symptomology, functioning and quality of life.
Time Frame: Baseline, 3 Months, 6 Months, 9 Months, 12 Months
Population: Deviations from in the number of participants result from missed visits, assessments and early exits.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Neurovascular Bundles and/or Urethra Included in Treatment: For patient self-completed assessments subjects were separated into two groups after the treatment (not randomly): 1) This group, neurovascular bundles and/or urethra included in treatment (n=57) or 2) Neurovascular bundles and urethra NOT included in treatment. There was no hypothesis test comparison. Comparisons are only observational. Deviations from the Overall Number of Participants is a result of missed visits, assessments and early exits.
- Neurovascular Bundles and Urethra Not Included in Treatment: For patient self-completed assessments subjects were separated into two groups after the treatment (not randomly): 1) Neurovascular bundles and/or urethra included in treatment (n=57) or 2) This group, neurovascular bundles and urethra NOT included in treatment. There was no hypothesis test comparison. Comparisons are only observational. Deviations from the Overall Number of Participants is a result of missed visits, assessments and early exits.
- Total Exablate MR Guided Focus Ultrasound: Combined Groups: Exablate MR Guided Focused Ultrasound - Local treatment of prostate lesions using Magnetic Resonance guided focused ultrasound energy. Combined groups (n=101): 1) Neurovascular bundles and/or urethra included in treatment (n=57) or 2) Neurovascular bundles and urethra NOT included in treatment (n=44) after the treatment (not randomly).
Arm/Group | Neurovascular Bundles and/or Urethra Included in Treatment | Neurovascular Bundles and Urethra Not Included in Treatment | Total Exablate MR Guided Focus Ultrasound
Number analyzed (Participants) | 57 | 44 | 101
score on a scale
  Baseline: number analyzed (Participants) | 56 | 43 | 99
  Baseline | 134.2 (15.7) | 134.3 (11.6) | 134.2 (14.0)
  3 Months: number analyzed (Participants) | 56 | 44 | 100
  3 Months | 134.3 (13.2) | 127.8 (16.3) | 131.4 (14.9)
  6 Months: number analyzed (Participants) | 55 | 42 | 97
  6 Months | 132.4 (15.8) | 130.5 (12.9) | 131.6 (14.6)
  9 Months: number analyzed (Participants) | 50 | 38 | 88
  9 Months | 136.6 (12.5) | 129.2 (14.5) | 137.7 (13.4)
  12 Months: number analyzed (Participants) | 57 | 44 | 90
  12 Months | 134.6 (14.9) | 130.7 (13.0) | 132.9 (14.2)

8. Secondary Outcome: Functional Assessment of Cancer Therapy - Prostate (Fact-P) Trial Outcomes Index (TOI)
Description: Functional Assessment of Cancer Therapy - P (Fact-P) Trial Outcomes Index (TOI, Score range: 1-104). An alternative scoring method to the Fact-G Total is the Trial Outcome Index (TOI), which is the sum of the Physical, Functional, and Lung Cancer Subscales. The TOI is reported to be an efficient and precise summary index of physical and functional outcomes. Higher scores indicate less symptomology and better physical and functional outcomes.
Time Frame: Baseline, 3 Months, 6 Months, 9 Months, 12 Months.
Population: Deviations in sample size across visits are due to subjects missing visits, missing assessments, or exiting the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Neurovascular Bundles and/or Urethra Included in Treatment: For patient self-completed assessments subjects were separated into two groups after the treatment (not randomly): 1) This group, neurovascular bundles and/or urethra included in treatment (n=57) or 2) Neurovascular bundles and urethra NOT included in treatment). There was no hypothesis test comparison. Comparisons are only observational.
- Neurovascular Bundles and Urethra Not Included in Treatment: For self-completed assessments subjects were separated into two groups after the treatment (not randomly): 1) Neurovascular bundles and/or urethra included in treatment (n=57) or 2) This group, neurovascular bundles and urethra NOT included in treatment. There was no hypothesis test comparison. Comparisons are only observational.
- Total Exablate MR Guided Focus Ultrasound: Combined groups: Exablate MR Guided Focused Ultrasound - Local treatment of prostate lesions using Magnetic Resonance guided focused ultrasound energy. Combined groups (n=101)
Arm/Group | Neurovascular Bundles and/or Urethra Included in Treatment | Neurovascular Bundles and Urethra Not Included in Treatment | Total Exablate MR Guided Focus Ultrasound
Number analyzed (Participants) | 57 | 44 | 101
score on a scale
  Baseline: number analyzed (Participants) | 56 | 43 | 99
  Baseline | 89.9 (10.5) | 90.8 (7.6) | 90.3 (9.3)
  3 Months: number analyzed (Participants) | 56 | 44 | 100
  3 Months | 89.1 (10.2) | 86.0 (10.2) | 87.7 (10.3)
  6 Months: number analyzed (Participants) | 55 | 43 | 98
  6 Months | 88.8 (11.4) | 86.9 (9.1) | 88.0 (10.4)
  9 Months: number analyzed (Participants) | 50 | 38 | 88
  9 Months | 90.5 (9.8) | 86.4 (9.5) | 88.7 (9.9)
  12 Months: number analyzed (Participants) | 51 | 39 | 90
  12 Months | 89.9 (9.7) | 87.7 (8.0) | 88.9 (9.0)

9. Secondary Outcome: International Consultation on Incontinence Questionnaire (ICIQ-SF). Urinary Incontinence (ICIQ) Total Score
Description: Urinary incontinence (ICIQ) Total Score (Score range: 0-21) is a simple questionnaire for evaluating the frequency, severity, and impact of urinary incontinence. High scores indicate greater impairment. Lower scores indicate better outcomes. This questionnaire assesses urinary incontinence and its impact on quality of life (QoL). So, a lower score implies less frequent and less severe incontinence, which is generally considered favorable.
Time Frame: Baseline, 3 Months, 6 Months, 9 Months, 12 Months.
Population: Deviations from the overall number of participants are a result of missed visits, missed incomplete assessments, and early study exits
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Neurovascular Bundles and/or Urethra Included in Treatment: For patient self-completed assessments subjects were separated into two groups after the treatment (not randomly): 1) This group, neurovascular bundles and/or urethra included in treatment (n=57) or 2) Neurovascular bundles and urethra NOT included in treatment. There was no hypothesis test comparison. Comparisons are only observational.
- Neurovascular Bundles and Urethra Not Included in Treatment: For patient self-completed assessments subjects were separated into groups after the treatment (not randomly): 1) Neurovascular bundles and/or urethra included in treatment (n=57) or 2) This group, neurovascular bundles and urethra NOT included in treatment. There was no hypothesis test comparison. Comparisons are only observational.
- Total Exablate MR Guided Focus Ultrasound: Combined groups: Exablate MR Guided Focused Ultrasound - Local treatment of prostate lesions using Magnetic Resonance guided focused ultrasound energy, combined groups (n=101)
Arm/Group | Neurovascular Bundles and/or Urethra Included in Treatment | Neurovascular Bundles and Urethra Not Included in Treatment | Total Exablate MR Guided Focus Ultrasound
Number analyzed (Participants) | 57 | 44 | 101
score on a scale
  Baseline | 1.2 (2.2) | 1.5 (2.8) | 1.3 (2.5)
  3 Months: number analyzed (Participants) | 56 | 43 | 99
  3 Months | 2.0 (3.0) | 2.2 (2.7) | 2.1 (2.9)
  6 Months | 2.2 (3.1) | 2.0 (2.6) | 2.1 (2.9)
  9 Months: number analyzed (Participants) | 51 | 39 | 90
  9 Months | 2.0 (2.6) | 2.1 (2.7) | 2.0 (2.6)
  12 Months: number analyzed (Participants) | 51 | 39 | 90
  12 Months | 2.0 (2.8) | 1.8 (2.4) | 1.9 (2.6)

10. Secondary Outcome: International Prostate Symptom Score (IPSS Total Score)
Description: High scores indicate worse symptomology. The total I-PSS score can range from 0 (asymptomatic) to 35 (very symptomatic). Additionally, there's a question about quality of life due to urinary symptoms, where patients rate their feelings from "delighted" to "terrible" regarding their current condition. This assessment helps clinicians understand the severity of BPH symptoms and guide treatment decisions.
Time Frame: Baseline, 3 Months, 6 Months, 9 Months, 12 Months.
Population: Deviations from the Overall Number of Participants Analyzed resulted from missed visits, missed assessments or early study exits.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Neurovascular Bundles and Urethra Not Included in Treatment: For patient self-completed assessments subjects were separated into twe groups after the treatment (not randomly): 1) Neurovascular bundles and/or urethra included in treatment (n=57) or 2) This group, neurovascular bundles and urethra NOT included in treatment. There was no hypothesis test comparison. Comparisons are only observational.
Arm/Group | Neurovascular Bundles and/or Urethra Included in Treatment | Neurovascular Bundles and Urethra Not Included in Treatment | Total Exablate MR Guided Focus Ultrasound
Number analyzed (Participants) | 57 | 44 | 101
score on a scale
  Baseline | 8.5 (6.4) | 8.8 (6.0) | 8.6 (6.2)
  3 Months: number analyzed (Participants) | 56 | 41 | 97
  3 Months | 8.1 (6.5) | 8.1 (5.2) | 8.1 (6.0)
  6 Months: number analyzed (Participants) | 55 | 43 | 98
  6 Months | 7.5 (6.5) | 8.4 (5.8) | 7.9 (6.2)
  9 Months: number analyzed (Participants) | 55 | 43 | 90
  9 Months | 7.5 (5.6) | 8.4 (5.8) | 8.2 (6.0)
  12 Months: number analyzed (Participants) | 50 | 39 | 89
  12 Months | 7.6 (5.8) | 8.9 (6.4) | 8.2 (6.1)

11. Secondary Outcome: International Prostate Symptom Score (IPSS) - Quality of Life Score
Description: IPSS Urinary Symptoms (IPSS-QoL Score range: 0-5). Question 7 of the IPSS, the Quality-of-Life question, is "7. Nocturia: How many times do you typically get up at night to urinate? (Select from 0 to 5)." Zero (0) suggests no interference with sleep and 5 suggests greater interference with sleep. Thus, high scores indicate worse quality of life.
Time Frame: Baseline, 3 Months, 6 Months, 9 Months, 12 Months.
Population: Deviations from the overall number of participants result from missed visits, missed assessments, and early study exits.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Neurovascular Bundles and Urethra Not Included in Treatment: For patient self-completed assessments subjects were separated into two groups after the treatment (not randomly): 1) Neurovascular bundles and/or urethra included in treatment (n=57) or 2) This group, Neurovascular bundles and urethra NOT included in treatment. There was no hypothesis test comparison. Comparisons are only observational.
Arm/Group | Neurovascular Bundles and/or Urethra Included in Treatment | Neurovascular Bundles and Urethra Not Included in Treatment | Total Exablate MR Guided Focus Ultrasound
Number analyzed (Participants) | 57 | 44 | 101
score on a scale
  Baseline | 1.9 (1.5) | 1.6 (1.2) | 1.8 (1.4)
  3 Months: number analyzed (Participants) | 56 | 42 | 98
  3 Months | 1.2 (1.2) | 1.5 (1.2) | 1.3 (1.2)
  6 Months: number analyzed (Participants) | 56 | 43 | 99
  6 Months | 1.2 (1.1) | 1.3 (1.0) | 1.2 (1.1)
  9 Months: number analyzed (Participants) | 51 | 39 | 90
  9 Months | 1.1 (1.1) | 1.4 (1.0) | 1.2 (1.1)
  12 Months: number analyzed (Participants) | 50 | 39 | 89
  12 Months | 1.1 (1.0) | 1.4 (1.0) | 1.2 (1.0)

12. Secondary Outcome: International Index of Erectile Function (IIEF-15) Erectile Dysfunction Overall Satisfaction
Description: IIEF-15 Erectile Dysfunction Overall Satisfaction (IIEF-15 Overall Satisfaction range: 0-10). Low scores are worse.
Time Frame: Baseline, 3 Months, 6 Months, 9 Months, 12 Months.
Population: Deviations from the Overall Number of Participants Analyzed results from missed visits, missed or incomplete assessments, or early study exits.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Neurovascular Bundles and/or Urethra Included in Treatment | Neurovascular Bundles and Urethra Not Included in Treatment | Total Exablate MR Guided Focus Ultrasound
Number analyzed (Participants) | 57 | 44 | 101
score on a scale
  Baseline: number analyzed (Participants) | 55 | 44 | 99
  Baseline | 7.8 (2.3) | 7.0 (2.7) | 7.4 (2.5)
  3 Months: number analyzed (Participants) | 51 | 40 | 97
  3 Months | 6.8 (2.7) | 6.5 (2.5) | 6.7 (2.6)
  6 Months: number analyzed (Participants) | 53 | 38 | 95
  6 Months | 7.0 (2.7) | 6.9 (2.8) | 7.0 (2.7)
  9 Months: number analyzed (Participants) | 47 | 36 | 85
  9 Months | 6.9 (2.4) | 6.7 (2.5) | 6.8 (2.4)
  12 Months: number analyzed (Participants) | 47 | 36 | 85
  12 Months | 6.9 (2.5) | 7.3 (2.4) | 7.1 (2.5)

ADVERSE EVENTS:
Time Frame: Safety of Exablate prostate treatment will be collected for one year after Exablate
Groups:
- Exablate MR Guided Focus Ultrasound Treatment of Localized Intermediate Risk Prostate Lesions: Exablate MR Guided Focused Ultrasound for the local treatment of prostate lesions using Magnetic Resonance guided focused ultrasound energy
Arm/Group | Exablate MR Guided Focus Ultrasound Treatment of Localized Intermediate Risk Prostate Lesions
All-Cause Mortality (participants affected / at risk) | 0/101
Serious Adverse Events (participants affected / at risk) | 0/101
Other Adverse Events (participants affected / at risk) | 24/101
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exablate MR Guided Focus Ultrasound Treatment of Localized Intermediate Risk Prostate Lesions (N=101)
Hematuria (Renal and urinary disorders) | 24 (25)
Urinary Incontinence (Renal and urinary disorders) | 19 (21)
Erectile Dysfunction (Reproductive system and breast disorders) | 19 (19)
Urinary Retention (Renal and urinary disorders) | 15 (17)
Penile / Testicular Pain (Reproductive system and breast disorders) | 14 (15)
Hematospermia (Reproductive system and breast disorders) | 13 (13)
Fatigue (General disorders) | 9 (10)
Ejaculation Disorder (Reproductive system and breast disorders) | 9 (9)
Urinary Frequency (Renal and urinary disorders) | 9 (9)
Urinary Tract Pain (Renal and urinary disorders) | 6 (6)
Urinary Hesitancy (Renal and urinary disorders) | 6 (6)
Urinary Urgency (Renal and urinary disorders) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI needs to consult Sponsor for accuracy of trial results and approval before being published

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-24): https://cdn.clinicaltrials.gov/large-docs/42/NCT01657942/Prot_SAP_000.pdf